CLINICAL TRIAL: NCT04470505
Title: Optimizing Platelet Isolation for Measures of Human Platelet Mitochondrial Respiration (The Cell Study)
Brief Title: Optimizing Platelet Isolation (The Cell Study)
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 260236
Record Dates: First submitted 2020-07-02; First posted 2020-07-14 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The research study is about blood cells (platelets) and their power houses (mitochondria). The investigators want to learn about their behavior in order to ensure that our laboratory procedures are generating optimal results.

DETAILED DESCRIPTION:
The objectives of this study are to assess platelet activation following standard laboratory procedures used in the process of measuring platelet mitochondrial function, and to determine the optimal amount of digitonin needed to permeabilize platelet cell membrane.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-35
* All races
* All ethnicity
* 18.5 - 30 BMI

Exclusion Criteria:

* smoking
* Aspirin intake
* Recreational drug use
* Alcohol intake more than 3 times per week
* Self-reported possibility of current pregnancy
* Known diagnosis of:
* Pre-diabetes
* Diabetes
* High cholesterol
* High triglycerides
* Hypertension
* Anemia
* Autism spectrum disorder
* Attention deficit hyperactivity disorder (ADHD)
* Attention deficit disorder (ADD)
* Severe asthma
* Refusal to stop taking nutritional supplements
* Any other pre-existing medical condition that requires daily medication as determined by the investigators to affect outcome of interest

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 25-35 years old
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Platelet activation from isolated platelets | day 1
  Whole blood will be collected following an overnight fast, and platelets isolated using standard procedures. Platelet activation markers (e.g., CD62P ) will be measured using flow cytometric analysis.

SECONDARY OUTCOMES:
Platelet activation measured in whole blood | day 1
  Whole blood will be collected following an overnight fast. Platelet activation will be measured in whole blood by the expression CD62P
Platelet reactivity measured in whole blood | day 1
  Whole blood will be collected following an overnight fast. Platelet reactivity will be measured in whole blood with adenosine diphosphate (ADP).

CONTACTS AND LOCATIONS:
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States